CLINICAL TRIAL: NCT01272934
Title: A Randomized, Double-blind, Multi-center, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Diclofenac Sodium Topical Gel (DSG) 1% Applied Four Times Daily in Subjects With Acute Ankle Sprain
Brief Title: Efficacy and Safety of Diclofenac Sodium Topical Gel 1% Applied Four Times Daily in Subjects With Acute Ankle Sprain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VOSG-P-318
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Results first posted 2013-01-15 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Acute Ankle Sprain
Keywords: Ankle Sprain, soft tissue injury
MeSH Terms: conditions — Ankle Injuries; Soft Tissue Injuries | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Diclofenac sodium topical gel 1% (Experimental): Diclofenac sodium topical gel 1%
  Interventions: Drug: Diclofenac Sodium

INTERVENTIONS:
Drug: Diclofenac Sodium — Topical gel 1%-4 times daily
  Arms: Diclofenac sodium topical gel 1%
Other: Placebo — Topical gel-4 times daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of DSG 1% compared with placebo applied four times a day in subjects with acute ankle sprains under 'in-use' conditions, in particular with regard to pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years and over.Acute sprain of the lateral ankle, Grade I-II, meeting baseline pain intensity level. Injury within past 12 hours.

Exclusion Criteria:

* Pain medication was taken within the 6 hours that precede randomization.During the past 3 months: Grade I-III sprain of the same ankle.During the past 6 months: Grade II-III sprain, any other significant injury (such as fracture or torn ligament), or surgery (except for skin or nails) of the same ankle or foot.Pain or instability in the same ankle attributable to previous ankle sprain or any other trauma.Ankle sprain attributable to a known disease affecting the ligaments, such as ligament hyperlaxity due to connective tissue disease (e.g., Marfan's syndrome, Down's syndrome, Ehlers-Danlos syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - NCH investigative site, Bad Nauheim
  - NCH investigative site, Brühl
  - NCH investigative site, Cologne
  - NCH investigative site, Essen
  - NCH investigative site, Gilching
  - NCH investigative site, Munich, Germany., Munich

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Start 18 January 2011 Study end 23 August 2011
Groups:
- Diclofenac Sodium Topical Gel 1%: Diclofenac sodium topical gel 1%
  Diclofenac Sodium : Topical gel 1%-4 times daily
- Placebo: Placebo : Topical gel-4 times daily
Period: Overall Study
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo
Started | 102 | 103
Completed | 102 | 101
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Abnormal Laboratory Value | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo | Total
Number analyzed (Participants) | 102 | 103 | 205
Age Continuous [Mean (Standard Deviation); unit: years] — Age : 18 years and over
  years | 32.5 (12.0) | 30.5 (10.8) | 31.5 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 55 | 104
  Male | 53 | 48 | 101
Region of Enrollment [Number; unit: participants]
  Germany | 102 | 103 | 205

OUTCOME MEASURES:

1. Primary Outcome: Pain on Movement
Description: Pain on Movement at 72 hours assessed on a 100 mm visual analog scale with anchors at 0="No pain" and 100= "Extreme pain"
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo
Number analyzed (Participants) | 102 | 103
mm | 25.6 (15.9) | 61.2 (16.6)

2. Secondary Outcome: Onset of Pain Relief
Description: Onset of perceptible pain relief.
Time Frame: On day 1
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo
Number analyzed (Participants) | 102 | 103
Hours | 4 [2 to 6] | NA [NA to NA] — Onset of Pain relief was not achieved for the first quartile within the given time frame in the placebo group

ADVERSE EVENTS:
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo
Serious Adverse Events (participants affected / at risk) | 0/102 | 1/103
Other Adverse Events (participants affected / at risk) | 6/102 | 3/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Sodium Topical Gel 1% (N=102) | Placebo (N=103)
Distorsion of wrist and ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Sodium Topical Gel 1% (N=102) | Placebo (N=103)
Infections and infestations (Infections and infestations) | 3 (3) | 2 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatobiliary disorders (Hepatobiliary disorders) | 0 (0) | 1 (1)
Nervous system disorders (Nervous system disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Preliminary agreement between Novartis Consumer Health and the investigator